CLINICAL TRIAL: NCT06774443
Title: Sensitivity of the Hinting Task in Patients With Huntington's Disease
Brief Title: Hinting Task for Huntington's Disease
Acronym: HT-HD
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: t.b.a
Record Dates: First submitted 2024-12-03; First posted 2025-01-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Huntington Disease
Keywords: Social Cognition; Theory of Mind; Hinting Task; Huntington; CAG repeat
MeSH Terms: conditions — Huntington Disease | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HD: Will undergo a neuropsychological assessment
  Interventions: Other: Neuropsychological assessment

INTERVENTIONS:
Other: Neuropsychological assessment — Neuropsychological assessment consisting of tests measuring social cognition and memory

SUMMARY:
Huntington's disease (HD) is an autosomal dominant neurodegenerative disorder, characterized by movement disorders, behavioural disorders and cognitive decline. Especially the behavioural and cognitive symptoms of the disease lead to significant disability and burden for patients as well as caregivers. One of the cognitive domains affected by HD is social cognition. Social cognition is the ability to perceive, interpret and respond correctly to social information. Aspects of social cognition are emotion recognition, perspective taking (Theory of Mind), and emapathy. Social cognition problems can be related to behavioural problems, but to be able to study this relationship, it is important to be able to reliable measure social cognition impairments. There are a few social cognition tests available, but often they are not normd and validated for use in a Dutch neurological population. There is a lack of sensitive, simple, tests for measuring Theory of Mind in patients with HD. A promising test, that already has been proven valid in a psychiatric population, is the Hinting Task. The Hinting Task measures theory of mind through indirect speech, The Hinting task is a social cognition test, where hints are implicitly given in speech, which resembles what patients and caregivers frequently report as difficult in HD. The Hinting Task has already been translated into Dutch and is already being used in clinical parctice, but its sensitivity has not been studied yet in a neurological population. The aim of this study is to assess if the Hinting Task is sensitive in patients with HD and to relate the Hinting Task to other (social) cognitive measures, demographical characteristics and disease characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Huntington's disease via CAG-repeat length analysis, minimum of 40 repeats
* Between 18 and 74 years of age
* Dutch speaking

Exclusion Criteria:

* Presence of serious psychiatric disorders or other neurological comorbidities

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We aim to include 47 patients with premanifest HD and 20 patients with manifest HD. Patients will be recruited from the Enroll-HD sample of the UMCG and the Huntington outpatient clinic of Noorderbreedte in Grou. All stuParticipants of Enroll-HD that have given consent to be asked to take part in other studies of HD, will be asked to participate in the current study. The study will also be advertised on the website of the Dutch Huntington Society. Participants can sign themselves up via that advertisement. Inclusion and all other study-related activities will be performed by UMCG study staff.
  Data of healthy controls on the Hinting Task has already been obtained from previous studies, and can be used in accordance with the FAIR data principles. Data of healthy controls that have given permission to use their data in similar studies will be included. Controls will be matched to patients so that sex and age distributions do not significantly differ between groups.
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance on the Hinting Task | 2025-2026
  Performance on the Hinting Task by patients with Huntington's disease compared to healthy controls

SECONDARY OUTCOMES:
Relations of the Hinting Task with other variables | 2025-2026
  Relationship of the Hinting Task with other (social) cognitive tests, disease characteristics and demographical characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Maraike Coenen, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared upon request.